CLINICAL TRIAL: NCT01745549
Title: Efficacy, Safety and Satisfaction of the New Pen Needle 33G x 4 mm 33G x 4 mm: Cross-over Randomized Controlled Clinical Trial. Studio AGO 01
Brief Title: Efficacy, Safety and Satisfaction of the New Pen Needle 33 Gauge x 4 mm.
Acronym: AGO01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorzio Mario Negri Sud (Other)
Collaborators: Artsana SpA (Unknown)
Responsible Party: Principal Investigator, Antonio Nicolucci, Dr Antonio Nicolucci, MD, Consorzio Mario Negri Sud
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AGO01
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: diabetes; insulin therapy; needle
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- needle 4 mm gauge 33 (Experimental): Needle for insulin pen, 4 mm long and with a diameter of 33 gauge (the smaller needle)
  Interventions: Device: Needle for insulin pen, 4 mm long and with a diameter of 33 gauge
- needle 4 mm gauge 32 (Active Comparator): Needle for insulin pen, 4 mm long and with a diameter of 32 gauge
  Interventions: Device: Needle for insulin pen, 4 mm long and with a diameter of 32 gauge

INTERVENTIONS:
Device: Needle for insulin pen, 4 mm long and with a diameter of 33 gauge
  Arms: needle 4 mm gauge 33
Device: Needle for insulin pen, 4 mm long and with a diameter of 32 gauge
  Arms: needle 4 mm gauge 32

SUMMARY:
During the last years, even more little needles are used for the injection of sub cutaneous insulin, for the diabetes therapy.

The aim of this study is to evaluate the non inferiority of a new needle, smaller than another needle, in terms of hematic levels od fructosamine, an indicator of glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 or type 2 diabetes
* both males and females
* age >=18 anni
* insulin treatment from at least 6 months
* signed informed consent

Exclusion Criteria:

* pregnancy
* incapacity for filling in the questionnaires
* every illness or condition that, according to the investigator, could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
hematic fructosamine levels | Change from baseline in fructosamine levels after 3 weeks of treatment

SECONDARY OUTCOMES:
mean amplitude of glucose excursions (MAGE) | Change from baseline in MAGE after 3 weeks of treatment
pain | questionnaire at the end of the treatments (at 6 weeks)
  visual analogic scale (VAS) 1-10
leakage at the site injection | number of episodes of leakage during the treatment (3 weeks)
  visual scale
hypoglycemia | number of episodes of hypoglycemia during the treatment (3 weeks)
insulin dosage | Change from baseline in insulin dosage after 3 weeks of treatment
patient's weight | Change from baseline in weight after 3 weeks of treatment
patient's satisfaction | questionnaire at the end of the treatments (at 6 weeks)
  VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nicolucci, MD, Study Chair — Consorzio Mario Negri Sud
Locations (4):
- Italy (4):
  - UO Malattie Metaboliche e Diabetologia - Ospedale di Treviglio-Caravaggio, Treviglio, BG
  - UO Diabetologia per Trattamento e Educazione dei Diabetici - Spedali Civili di Brescia, Brescia, BS
  - U.O.S. Diabetologia e Malattie Metaboliche - PO Cantù - Mariano Comense, Mariano Comense, CO
  - Struttura Complessa Dietologia-Diabetologia Malattie Metaboliche - Ospedale Pertini, Roma, RM

REFERENCES:
- [Derived] Valentini M, Scardapane M, Bondanini F, Bossi A, Colatrella A, Girelli A, Ciucci A, Leotta S, Minotti E, Pasotti F, Pesenti A, Rocca L, Sciangula L, Vavassori E, Nicolucci A. Efficacy, safety and acceptability of the new pen needle 33G x 4 mm. AGO 01 study. Curr Med Res Opin. 2015 Mar;31(3):487-92. doi: 10.1185/03007995.2014.993025. Epub 2014 Dec 10. PMID 25469829